CLINICAL TRIAL: NCT03945097
Title: University of Washington Reading & Dyslexia Research Program
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jason Yeatman, Assistant Professor, Institute for Learning & Brain Sciences, Dept. of Speech & Hearing Services, University of Washington
Other Study IDs: STUDY00000516; 1R21HD092771-01A1 (NIH)
Record Dates: First submitted 2019-04-26; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Reading Disability
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Letters: Education program focuses on learning letters.
  Interventions: Behavioral: preK
- Language: Education program focuses on language comprehension.

INTERVENTIONS:
Behavioral: preK — Subjects enter and education program that either focuses on learning letters and their corresponding sounds or on language comprehension skills.
  Groups: Letters

SUMMARY:
Subjects are recruited for a pre-kindergarten education program focusing on early literacy skills. Primary outcomes are improvement in letter knowledge and changes in brain response to text.

ELIGIBILITY:
Inclusion Criteria: Typically developing children enrolled before kindergarten.

* Typically developing child between 60 and 72 months of age
* Has not yet begun Kindergarten

Exclusion Criteria:

* Reported neurological or psychiatric condition.
* Claustrophobia. ADHD

Ages: 60 Months to 72 Months | Sex: All
Age Groups: Child
Study Population: Typically developing children
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Letter Knowledge | Within 2 weeks post intervention
  Knowledge of letter names and sounds. This is computed as percent correct (out of 52). Each child is shown a flash card with each upper case letter and asked to name it and say its sound

CONTACTS AND LOCATIONS:
Overall Officials: Jason Yeatman, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washignton, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No